CLINICAL TRIAL: NCT04283955
Title: A Retrospective Cohort Study: The Influence of MTHFR C677T and A1298C on the High-dose Methotrexate-Related Toxicities in Pediatric Patients With Non-Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-Fei Sun, MD, Sun Yat-sen University
Other Study IDs: SCCCG-NHL-2017
Record Dates: First submitted 2020-02-23; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pediatric NHL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: High-dose MTX based chemotherapy — Patients received MTX therapy at the dose of 5g/m2 for 24 hours. Each dose of HD-MTX therapy was followed by 6~7 times of leucovorin rescue 12 hours after the end of MTX infusion, at the dose of 15 mg/ m2 every 6 hours. The plasma MTX levels were monitored at 0, 24, 48, 72 hours from the initiation of HD-MTX infusion. To maintain the urine pH at approximately 7~8, intravenous hydration and alkalization at the dose of 1,500ml/ m2 per day were achieved 12 hours prior to the initiation of HD-MTX administration (D0) and 3,000ml/ m2 per day lasted for the following 3 days (D1 to D3). CF was used to rinse mouth to prevent oral mucositis from D1 to D3. We closely monitored the volume and pH of the urine via routine test from D0 to D4.

SUMMARY:
We hypothesized that polymorphism MTHFR C677T and A1298C should be associated with HD-MTX-related toxicities in children with NHL. Therefore, we aimed to retrospectively explore their relationships in this analysis.

DETAILED DESCRIPTION:
INTRODUCTION: Non-Hodgkin lymphoma (NHL), the fourth most common malignancy across the pediatric age spectrum, is a heterogeneous group of lymphoid malignancies. In children, NHL comprises four main wide categories: lymphoblastic lymphoma (LBL), Burkitt lymphoma (BL), diffuse large B-cell lymphoma (DLBCL), and anaplastic large cell lymphoma (ALCL). The current overall survival rate of pediatric NHL exceeds 80% due to dramatic progress in developing risk-adapted curative therapy (1), in which methotrexate (MTX) plays a crucial part.

MTX is used to treat a variety of cancers. A high-dose MTX (HD-MTX) regimen, referred to the administration of a dosage ranging from 0.5g/m2 to 12.0g/m2 or even higher, is commonly used to treat childhood acute lymphoblastic leukemia (ALL), lymphoma and pediatric osteosarcoma. Despite its wide range of therapeutic efficacy, the toxicities of HD-MTX including reversible myelosuppression, nausea, vomiting, diarrhea, hepatotoxicity, nephrotoxicity, neurotoxicity, and particularly oral mucositis should not be neglected. Accumulating pharmacogenetic studies have revealed that polymorphisms of enzymes involved in folate pathway could lead to variability in response to MTX and HD-MTX-related toxicities in various malignancies. The most two extensively studied SNPs of MTHFR in relation to the toxicities of MTX are the C677T variant (Ala222Val, rs1801133) and A1298C variant (Glu 429Ala, rs1801131), both dampening the enzyme activity by 40-70%.

However, limited evidence is available in pediatric NHL, with results varying considerably in different studies. Therefore, the aim of this retrospective study was to evaluate the influence of C677T and A1298C polymorphisms on HD-MTX-related toxicities in children with NHL treated according to BFM-modified protocols.

PATIENTS & METHODS：We reviewed the medical records of all pediatric patients who were diagnosed as NHL and received HD-MTX-based chemotherapy at the dose of 5g/m2 in Sun Yat-sen University Cancer Center between March 2014 and March 2019. Data were analyzed by chi-square test.

ELIGIBILITY:
Inclusion Criteria: patients who were:

* Aged ≤ 18 years old；
* Diagnosed as the four main types of NHL, including lymphoblastic lymphoma (LBL), Burkitt's lymphoma (BL), anaplastic large cell lymphoma (ALCL), diffuse large B-cell lymphoma (DLBCL);
* Treated with HD-MTX therapy at the dose of 5g/m2;
* Genotyped by PCR following Sanger with respect to MTHFR C677T and A1298C
* With complete medical records.

Exclusion Criteria: patients who were:

* Aged >18 years old；
* Diagnosed as cancer types other than the four main types of NHL;
* Treated with no HD-MTX therapy or at the dose other than 5g/m2;
* Not genotyped by PCR following Sanger with respect to MTHFR C677T and A1298C
* With incomplete medical records .

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Age：≤ 18 years old；
  2. Diseases: the four main types of NHL, including lymphoblastic lymphoma (LBL), Burkitt's lymphoma (BL), anaplastic large cell lymphoma (ALCL), diffuse large B-cell lymphoma (DLBCL)
  3. Treatment: HD-MTX-based chemotherapy at the dose of 5g/m2;
  4. Genotype: MTHFR C677T and A1298C；
  5. Center：Sun Yat-sen University Cancer Center，Guangzhou, P.R China;
  6. Time period: between March 2014 and March 2019.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Observations of HD-MTX-related toxicities | 3 weeks
  We recorded the toxicities that occurred to the patients after the MTX infusion, including hematological suppression, hepatotoxicity, nephrotoxicity, oral mucositis, vomiting and diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China